CLINICAL TRIAL: NCT02393079
Title: The Effects of Transcranial LED Therapy (TCLT) in Patients With Traumatic Brain Injury (TBI): a Prospective, Randomized Controlled Trial
Brief Title: Analysis of TCLT in TBI Patients: a Prospective, Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Guilherme da Cruz Ribeiro Poiani, Principal Investigator - clinical neuropsychologist, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCLT/DIP
Record Dates: First submitted 2015-02-20; First posted 2015-03-19 (Estimated); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Brain Injury; Cognitive Deficits
Keywords: Traumatic Brain Injury; Cognitive
MeSH Terms: conditions — Brain Injuries; Cognition Disorders; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active helmet LED (Experimental): Description of the intervention: 18 patients will undergo 18 sessions of transcranial LED therapy (ACTIVE HELMET) with 30 minutes duration each. The sessions take place over 6 weeks. The therapy will be performed with a helmet that covers the frontal and parietal region.
  Interventions: Device: Transcranial LED Therapy (TCLT)
- Sham group (Sham Comparator): Description of the intervention: 18 patients will undergo 18 sessions of transcranial LED therapy (INACTIVE HELMET) with 30 minutes duration each. The sessions take place over 6 weeks. The therapy will be performed with a helmet that covers the frontal and parietal region.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Transcranial LED Therapy (TCLT) — Whereas the geometry of the skull and to uniformly distribute the light radiation, the TLTC is applied using as light source a set of LEDs installed in a helmet, emitting radiation in the range between 600nm and 650nm with a peak at 630nm, so in the red region.
  Arms: Active helmet LED
Device: Sham — A SHAM identical helmet will be used in the control group.
  Arms: Sham group

SUMMARY:
The purpose of this study is to evaluate the early and late effects of Transcranial Led Therapy (TLTC) in memory and executive functions in patients with moderate and severe TBI history (TBI time longer than 3 months).

DETAILED DESCRIPTION:
In the current study patients in the outpatient center - Neurotrauma Unit at University of São Paulo (HCFMUSP) diagnosed with moderate / severe blunt head trauma that meet the inclusion criteria will be divided randomly and blindly in two groups: Group A (n = 18) will receive stimulation through active helmet and Group B (n = 18) given placebo stimulation or sham through the inactive helmet. All patients will be subjected to 3 times of neuropsychological assessment: Study 1 (E1) - up to 4 weeks before the start of TLTC sessions; Study 2 (E2) - a week after the end of TLTC; and Study 3 (E3) - three months after the intervention. The evaluations will take in order to verify the early and late effects of TLTC in attention, memory and executive functions in patients with moderate and severe TBI.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis of traumatic brain injury
* Must be able to sign the Informed Consent Form
* Patients with TBI beginning three months after injury

Exclusion Criteria:

* Impairment of language and / or limiting engine
* Extensive Cranial vault defects
* Presence of uncontrolled post-TBI epilepsy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-01; Primary Completion 2019-06 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Evidence of improvement in inhibitory control measured by cognitive assessment (Stroop Test - Victoria Version) in patients undergoing intervention with an active LED helmet. | Three times: Up to one week before to start intervention, one week and three months after end the intervention
  Measurement of each patient's inhibitory control by means of a test that causes them to cognitively suppress a habitual response in favor of a less habitual one. The results of patients with shorter response times indicate better positions in the tables, according to age. Examples of the average time (in seconds) of best results are between 17-29 years (11.79) and 80+ (19.31), any time longer than these indicates decreasing results.

SECONDARY OUTCOMES:
Assess the immediate and late effects of the intervention on victims of moderate or severe TBI in the following cognitive domains: executive functioning, attentional processes and memory. | Three times: Up to one week before to start intervention, one week and three months after end the intervention
  Apply a neuropsychological assessment battery focused on executive functioning, attentional processes and memory to measure the effects of the active led helmet compared to the use of the sham device.

CONTACTS AND LOCATIONS:
Overall Officials: Wellingson S Paiva, MD PhD, Principal Investigator — Clinics Hospital - University of Sao Paulo Medical School
Locations (1):
- Clinics Hospital - University of Sao Paulo Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Poiani GDCR, Zaninotto AL, Carneiro AMC, Zangaro RA, Salgado ASI, Parreira RB, de Andrade AF, Teixeira MJ, Paiva WS. Photobiomodulation using low-level laser therapy (LLLT) for patients with chronic traumatic brain injury: a randomized controlled trial study protocol. Trials. 2018 Jan 8;19(1):17. doi: 10.1186/s13063-017-2414-5. PMID 29310710